CLINICAL TRIAL: NCT06921174
Title: Comparison of the Effectiveness of Classical Perineal Massage Therapy Versus the Use of an Intravaginal Device to Reduce Postpartum Perineal Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Sexológico Murciano (Other)
Collaborators: CIAGO - Center for Comprehensive Gynecology and Obstetrics (Unknown); Carmen Parra Pilates Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.P. ISM-CRE-2024-01
Record Dates: First submitted 2025-03-27; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Pelvic Pain
Keywords: postpartum pelvic pain
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Intervention Model Description: Type: Randomized Controlled Trial (RCT)
  Structure: Two parallel groups (random assignment)
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Classical Perineal Massage Therapy (Active Comparator): Performed manually by a pelvic floor physiotherapist.
  One 30-minute session per week for 12 weeks.
  Interventions: Procedure: Classical Perineal Massage Therapy
- Use of the "Crescendo 2" Intravaginal Device (Experimental): Self-administered perineal massage at home.
  Three times per week, 10 minutes each session, over a 12-week period.
  Interventions: Device: Use of the "Crescendo 2" Intravaginal Device

INTERVENTIONS:
Device: Use of the "Crescendo 2" Intravaginal Device — Self-administered perineal massage at home with Crescendo device.
  Three times per week, 10 minutes each session, over a 12-week period.
  Arms: Use of the "Crescendo 2" Intravaginal Device
Procedure: Classical Perineal Massage Therapy — Performed manually by a pelvic floor physiotherapist.
  One 30-minute session per week for 12 weeks.
  Arms: Classical Perineal Massage Therapy

SUMMARY:
GA34.01 postpartum, a randomized design with a parallel group structure will be applied, randomly assigning participants into two groups. The first group will receive the traditional perineal massage therapy, while the second group will use the intravaginal device "Crescendo 2." In this study, a pre- and post-intervention evaluation will be conducted, using the Visual Analog Scale (VAS) as the primary outcome measure and the Clinical Global Impression Scale as the secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older.
* Residing in the Region of Murcia.
* Having had a vaginal delivery between 6 weeks and 12 months prior to enrollment.
* Presenting postpartum perineal pain, coded in ICD-11 as GA34.01.
* Have not received any prior treatment for this condition.

Exclusion Criteria:

* Presence of severe conditions such as:
* Excessive postpartum hemorrhage
* Serious infections
* Respiratory or circulatory complications
* Neurological disorders requiring intensive medical intervention
* Currently under pharmacological treatment for pelvic pain.
* Active vaginal infections.
* Expressed refusal to participate or inability to comply with study procedures.
* Women with episiotomy may participate only if there were no complications such as severe infection or hemorrhage following the procedure.

Willingness to participate and to follow the study protocol.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) - to assess pain intensity | First measure week 1 and Last measure week 12
  The **Visual Analogue Scale (VAS)** will be used as the **primary outcome measure**. It consists of a horizontal line approximately 10 centimeters long. At each end of the line are the extreme expressions of pain: on the left, "no pain," and on the right, "worst imaginable pain." This tool allows us to measure the intensity of pain with high reproducibility between observers.
  Visual Analogue Scale (VAS):
  The Visual Analogue Scale is a psychometric response scale used to measure pain intensity. It typically consists of a 10-centimeter horizontal line anchored by two verbal descriptors: "no pain" (score = 0) and "worst imaginable pain" (score = 10).
  Minimum score: 0 (no pain) Maximum score: 10 (worst imaginable pain) Interpretation: Higher scores indicate worse outcomes (i.e., more intense pain).

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) - for overall health status | At the end of the treatment week 12
  The Clinical Global Impression Scale (CGI) will be used as the secondary outcome measure.
  The Global Impression Scale (GIC) is a subjective tool used to assess the overall perceived change in a patient's health status, particularly in clinical studies involving various conditions and treatments.
  Clinical Global Impression - Change (CGI-C) Scale:
  The Clinical Global Impression - Change scale is a clinician-rated tool used to assess changes in a patient's condition over time, relative to baseline.
  Minimum score: 1 (very much improved) Maximum score: 7 (very much worse) Interpretation: Lower scores indicate better outcomes (i.e., greater clinical improvement), while higher scores indicate worsening.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Sexológico Murciano, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schulz KF, Grimes DA. Generation of allocation sequences in randomised trials: chance, not choice. Lancet. 2002 Feb 9;359(9305):515-9. doi: 10.1016/S0140-6736(02)07683-3. PMID 11853818
- [Background] Beckmann MM, Garrett AJ. Antenatal perineal massage for reducing perineal trauma. Cochrane Database Syst Rev. 2006 Jan 25;(1):CD005123. doi: 10.1002/14651858.CD005123.pub2. PMID 16437520
- See also: Related Info — https://www.isemu.es
- Available data/document: Study Protocol — https://www.isemu.es